CLINICAL TRIAL: NCT06545097
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Cebranopadol for the Treatment of Moderate to Severe Acute Pain After Full Abdominoplasty
Brief Title: A Study of Cebranopadol for the Treatment of Acute Pain After Abdominoplasty
Acronym: ALLEVIATE1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRN-228-301
Record Dates: First submitted 2024-08-06; First posted 2024-08-09 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Acute Pain
Keywords: Abdominoplasty
MeSH Terms: conditions — Acute Pain | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Treatment A (Experimental): Cebranopadol 400 ug (once daily for 2 days)
  Interventions: Drug: Cebranopadol 400 ug
- Treatment B (Experimental): Cebranopadol 400 ug on Day 1; 200 ug on Day 2
  Interventions: Drug: Cebranopadol 400 ug; Drug: Cebranopadol 200 ug
- Treatment C (Placebo Comparator): Placebo (once daily for 2 days)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cebranopadol 400 ug — Once daily
  Other Names: TRN-228
  Arms: Treatment A; Treatment B
Drug: Cebranopadol 200 ug — Once daily on Day 2
  Other Names: TRN-228
  Arms: Treatment B
Drug: Placebo — Once daily for 2 days
  Arms: Treatment C

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of Cebranopadol for acute pain after a Abdominoplasty.

DETAILED DESCRIPTION:
This study is a Phase 3, multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Cebranopadol for the Treatment of Moderate to Severe Acute Pain after Full Abdominoplasty. This study will be conducted in 3 phases: Screening, Treatment, and Follow-up.

ELIGIBILITY:
Key Inclusion Criteria:

* Scheduled to undergo full abdominoplasty procedure without liposuction or other collateral procedures, using anesthesiologic and surgical procedures planned as described in this protocol.
* Must be able to adhere to the visit schedule, complete all study assessments, and protocol requirements including self-reported questionnaires.

Key Exclusion Criteria:

* Any clinically significant disease, medical condition or laboratory finding that in the investigator's opinion may interfere with the study procedures or data integrity or compromise the safety of the subject.
* Subject has a current painful condition that could confound the interpretation of efficacy, safety or tolerability data in the study, in the opinion of the investigator.
* History of allergy, hypersensitivity or intolerance to any opioid analgesics or anesthetics, including opioid-induced nausea or vomiting.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 279 (Actual)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
Primary Outcome Measure | 4-48 hours
  Pain Numerical Rate Scale (NRS) area under the curve from 4 through 48 hours (AUC4-48)

SECONDARY OUTCOMES:
Secondary Outcome Measure: | 4-48 hours
  Pain Numerical Rate Scale (NRS) AUC4-24
Secondary Outcome Measure: | 48 hours
  Number of doses of rescue medication
Secondary Outcome Measure: | 24-48 hours
  Pain NRS AUC
Other Secondary Endpoint | Partial AUCs: 4-12, 12-24, 24-36, 36-48, and 4-36 hours
  Pain NRS
Other Secondary Endpoint | Proportion of subjects who take at least 1 dose of rescue medication up to hours 12, 24, and 36
  Rescue Medication
Other Secondary Endpoint | peak sedation, total score and AUC4-48
  MOAA/S

CONTACTS AND LOCATIONS:
Overall Officials: Harold S. Minkowitz, MD, Principal Investigator — HD Research
Locations (4):
- United States (4):
  - ALLEVIATE 1 Site 001106, Little Rock, Arkansas
  - ALLEVIATE 1 Site 001112, Miami, Florida
  - ALLEVIATE 1 Site 001110, Bellaire, Texas
  - ALLEVIATE 1 Site 001111, San Antonio, Texas